CLINICAL TRIAL: NCT06785116
Title: A Randomized, Placebo-controlled Trial of DAPAgliflozin for Cardiovascular Risk Reduction in the Postpartum Period of Hypertensive Pregnancies
Brief Title: A Randomized, Placebo-controlled Trial of DAPAgliflozin (DAPA) for Cardiovascular Risk Reduction in the Postpartum Period of Hypertensive Pregnancies (HP)
Acronym: DAPA-HP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Society for Maternal-Fetal Medicine Foundation (Unknown); American Association of Obstetricians and Gynecologists Foundation (Unknown)
Responsible Party: Principal Investigator, Ashley Hesson, Assistant Professor of Obstetrics and Gynecology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00260815
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Gestational Hypertension; Hypertension in Pregnancy; Pre-Eclampsia; Superimposed Pre-Eclampsia; Cardiovascular Complication
Keywords: Medication; Placebo; Postpartum period; Cardiovascular risk reduction; Echocardiogram
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: The study will be conducted in a 1:1 fashion between the DAPA Group and the Control Group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, the clinical team, and researchers will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Dapagliflozin (Experimental): 10 Milligram (mg) orally
  Interventions: Drug: Dapagliflozin 10mg Tab

INTERVENTIONS:
Drug: Placebo — Participants will take this daily for 6-months. Additionally, during the study participants will have 4 study visits and be asked to complete study specific activities (i.e. daily blood pressure, weekly weights, laboratory draws, echocardiograms, etc.) Participants will be followed remotely for 1-month after the 6-month visit.
  Arms: Placebo
Drug: Dapagliflozin 10mg Tab — Participants will take this daily for 6-months. Additionally, during the study participants will have 4 study visits and be asked to complete study specific activities (i.e. daily blood pressure, weekly weights, laboratory draws, echocardiograms, etc.) Participants will be followed remotely for 1-month after the 6-month visit.
  Other Names: Farxiga
  Arms: Dapagliflozin

SUMMARY:
This trial is a pilot-scale, single institution randomized, placebo-controlled trial to assess the feasibility, acceptability, and efficacy of administering dapagliflozin for cardiovascular risk reduction in the postpartum period. The target population is patients at high risk of adverse cardiovascular outcomes within five years post-delivery.

Eligible participants will be randomized to receive either: 1) dapagliflozin (10mg daily) for six months (DAPA group) or 2) an orally administered, daily placebo (Control group).

The study hypothesizes:

The dapagliflozin group will have higher cardiovascular risk reduction scores than the Control Group.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for delivery at the University of Michigan (UM) Labor and Delivery (L&D) unit or enrolled in the UM postpartum blood pressure monitoring program following a delivery at the UM L&D unit
* Determined to be at least 23 and 0/7 weeks of gestation based on a clinically acceptable dating method (can be a single or multifetal gestation with or without the presence of fetal anomalies) at the time of delivery
* Consents to participation and must understand/read/speak English with the ability to understand and willingness to sign a written informed consent in English
* Diagnosed with a hypertensive pregnancy by either of the following criteria:

  * Taking an antihypertensive medication for the diagnosis of chronic or essential hypertension at the time of admission
  * Hypertension, chronic hypertension, or essential hypertension must be present in the prospective participant's medical record
  * Antihypertensive" can be any medication taken for the purpose of blood pressure control per the medical record
  * A documented hypertensive disorder of pregnancy (gestational hypertension, preeclampsia without severe features, preeclampsia with severe features, superimposed preeclampsia, or eclampsia) prior to delivery
* Eligible participants must report a planned contraceptive method as part of the consent process, to be noted on their consent document.
* Has two or more blood pressures ≥160/110 Millimeters of mercury (mmHg) at least 60 minutes apart

  * If an admitted patient does not meet this blood pressure criterion but is otherwise eligible, participants can consent to have a BNP drawn within 12 hours of delivery as an alternative measure of cardiovascular risk (if the brain natriuretic peptide (BNP) is ≥100 Picograms per milliliter (pg/ml), participants are eligible to participate)

Exclusion Criteria:

* Non-English speaking
* Ongoing pregnancy
* Stated desire to become pregnant within 8 months post-delivery
* Intention to breastfeed after enrollment
* BNP ≥1000 pg/ml within 12 hours of delivery, clinical team to be notified of result
* Comorbidities that may affect cardiovascular risk assessment (per protocol)
* Contraindication to dapagliflozin (per protocol)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-02 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular risk reduction score | Baseline, 6 months
  The score will be summed and compared between groups.The components with outcome-based binary assessments by the following:
  * Biometric: change in systolic blood pressure (scores of 0 or 1) and change in body weight (scores of 0 or 1)
  * Echocardiogram: change in left ventricle wall thickness (scores of 0 or 1) and change in left ventricle mass (scores of 0 or 1)
  * Clinical: Non-hospitalization (scores of 0 or 1) and return to baseline antihypertensive needs (scores of 0 or 1) The total scores range from 0-6 with a higher score indicating greater cardiovascular risk reduction.

SECONDARY OUTCOMES:
The number of patients screened | 2-year recruitment period
The number of patients screen-outs vs screen-ins | 2-year recruitment period
  These will be the participants that qualify either by blood pressure or laboratory parameter (BNP) (screen-ins) or if not eligible (screen-outs).
Reasons for ineligibility and refusal to participate | 2-year recruitment period
Patient-stated adherence | baseline to 6 months
  This will be collected by the patient medication diary and study visit questionnaire.
Patient reported barriers to adherence | baseline to 6 months
  Participants will answer 2 questions regarding missed doses of medications. These will be summarized.
Loss to follow-up rates | Baseline to 6 months
  Information on loss to follow-up (where available) will be reported to inform future work.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Hesson, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No